CLINICAL TRIAL: NCT02827916
Title: Exploration of Neuropathic Pain Induced by Oxaliplatin Electrophysiological Approach: Interest Using the SUDOSCAN® Machine
Brief Title: Exploration of Neuropathic Pain Induced by Oxaliplatin Electrophysiological Approach
Acronym: CANALOXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CANALOXA
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Peripheric Neuropathy; Chemo-induced Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): Measure of painful neuropathy for al patients with thermotest and sudoscan Devices and Neuropathic Pain Symptom Inventory.
  Interventions: Device: Assessment of neuropathic pain with theThermotest device; Device: Assessment of neuropathic pain with SUDOSCAN device; Device: Assessment of neuropathic pain with the Neuropathic Pain Symptom Inventory.

INTERVENTIONS:
Device: Assessment of neuropathic pain with theThermotest device — Measure of painful neuropathy with thermotest
Device: Assessment of neuropathic pain with SUDOSCAN device — Measure of painful neuropathy with sudoscan Devices
Device: Assessment of neuropathic pain with the Neuropathic Pain Symptom Inventory. — Measure of painful neuropathy with Neuropathic Pain Symptom Inventory.

SUMMARY:
Oxaliplatin is an anticancer agent commonly used in the treatment of colorectal cancer. However, the development of neuropathic pain under treatment limits its use. These are manifested by acute hyperesthesia / distal cold allodynia and chronic course of hypoesthesia.

It is widely reported that these pains are consecutive to hyperexcitability of some ioniques2 channels (mainly sodium and potassium channels). However, the pathophysiological mechanisms of neurotoxicity are multifactorial and still imperfectly described.

Since May 2014, the hospital group Paris Saint Joseph led the pilot study LIPIDOXA whose challenge is to quantify / measure NAION and explained by a biochemical approach, specifically Lipidomics. The CANALOXA study is the logical continuation of LIPIDOXA study insofar design methodology relies heavily on techniques developed for LIPIDOXA study and that the expected results will be complementary to those of LIPIDOXA.

DETAILED DESCRIPTION:
Main objective:

it is, in cancer patients chronically treated with oxaliplatin (over 5 courses) and exhibiting signs of neuropathy, to correlate the quantitative changes in the thermal sensitivity to hot and cold (Thermotest, Quantitative Sensory Testing QST ) with any changes in the ion conductance chlorine measured by electrophysiological technique (SUDOSCAN).

Secondary objectives:

* Correlating the results obtained with both types of techniques and with the descriptive parameters of the population included.
* Understand the importance of regulating the activity of the chloride channel in the development of neuropathy induced by oxaliplatin.

Methodology :

Prospective study, single center, intervention in routine care. Time study: February 2015 - October 2016

1. Evaluation of neuropathy by electrophysiological methods (SUDOSCAN) The SUDOSCAN is a new technology fast and non-invasive to quantify the degree of neuropathy objectively through evaluation of chloride conductance at the skin of the palms and the soles of pieds4,5.
2. Evaluation of neuropathy by devices for quantitative measurement of neuropathic pain

   The pain symptoms was evaluated through various semi-objective neuropathy quantification tools (Quantitative Sensory Testing devices) 6:
   * The Thermotest (Somedic®): medical device that measures the thermal sensitivity thresholds to cold and hot: cold sensitivity threshold, threshold of sensitivity to hot, cold pain threshold, pain threshold warm. These stimuli are transmitted by the fiber Adelta and C. Since dysesthesia to thermal stimuli (allodynia in acute and chronical hypoesthesia) are typical of oxaliplatin, Thermotest is fundamental.
   * Questionnaire NPSI (Neuropathic Pain Symptom Inventory) widely used in the field and validated.
3. Statistical Analysis: Professor Gilles Chatellier, statistician (Clinical Research Unit, Hôpital Européen Georges Pompidou) will bring its expertise in statistical analysis.

NB: For each subject will be awarded an identifier (simple counter: increment as and measurement of inclusions) and the data will be entered on a computer file which will be sent to the statistician in charge of the analysis. There will be no exchange of personal data for this study is single center on the site GHPSJ.

Development of the study:

* Inclusion of patients treated with oxaliplatin from 6th cycle (FOLFOX protocols FOLFIRINOX, EOX, GEMOX, EOF, XELOX).
* Expected duration of patient recruitment: 9 months
* Number of patients to recruit and duration of participation for each patient: Based on 75 patients seen in 9 months in GHSPJ the oncology department for cancer of the digestive tract, and knowing that the prevalence of neuropathic pain in oxaliplatin is 50-70% (Attal 2009), the investigators plan to include at least 36 patients in this period of 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly treated with oxaliplatin
* Patient suffering from any type of cancer treated with oxaliplatin
* Man or Woman over 18

Exclusion Criteria:

* Patient with brain or leptomeningeal metastases
* Patient previously treated with cisplatin
* Patient addicted to alcohol
* Diabetic patient with peripheral neurological disorders
* Patient receiving calcium or magnesium salts intravenously
* Patient suffering from peripheral neuropathy
* Patient suffering from psychiatric disorders
* Patient treated with at least one of the following drug: venlafaxine, carbamazepine, gabapentin, pregabalin, clomipramine, amitriptyline, imipramine, duloxetine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of neuropathy by electrophysiological methods using SUDOSCAN | Day 1
  The SUDOSCAN is a new technology fast and non-invasive to quantify the degree of neuropathy objectively through evaluation of chloride conductance of the skin on the palm of the hand and soles of the feet2). This can evaluate the neuropathy for quantitative measurement of neuropathic pain

SECONDARY OUTCOMES:
Evaluation of neuropathy by devices for quantitative measurement of neuropathic pain | Day 1
  The pain symptoms are evaluated through various semi- objective neuropathy quantification tools (Quantitative Sensory Testing devices)6 :
  - Le Thermotest (Somedic®) : medical device that measures the thermal sensitivity thresholds to cold and hot: cold sensitivity threshold, threshold of sensitivity to hot, cold pain threshold, pain threshold warm. These stimuli are transmitted by the fiber Adelta and C. Since dysesthesia to thermal stimuli (allodynia in acute and hypoesthesia in chroniqe) are typical of oxaliplatin, Thermotest is fundamental.
NPSI ange of Characterization of pain neuropathy | Day 1
  Questionnaire NPSI (Neuropathic Pain Symptom Inventory) widely used in the field and validated.

CONTACTS AND LOCATIONS:
Overall Officials: COUDORE Francois, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Delmotte JB, Tutakhail A, Abdallah K, Reach P, D'Ussel M, Deplanque G, Beaussier H, Coudore F. Electrochemical Skin Conductance as a Marker of Painful Oxaliplatin-Induced Peripheral Neuropathy. Neurol Res Int. 2018 Sep 27;2018:1254602. doi: 10.1155/2018/1254602. eCollection 2018. PMID 30363900